CLINICAL TRIAL: NCT06341153
Title: The Effect of Breastmilk Smelling and Tasting & Smelling First Breastfeeding Practices on Sucking Success and Early Period Feeding Clues of Term Newborns
Brief Title: The Effect Of Breast Milk Sniffing And Tasting On Early Feeding Tips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Küçükoğlu (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor-Investigator, Sibel Küçükoğlu, Responsible researcher (Prof), Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SelcukUni2542
Record Dates: First submitted 2024-03-15; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Breastfeeding; Odors, Body; Newborn; Vitality
MeSH Terms: conditions — Breast Feeding; Body Odor | interventions — Taste

STUDY DESIGN:
Intervention Model Description: The stratification and blocking method was used to assign the mothers who would participate in the study to the experimental and control groups, taking into account factors such as normal or cesarean delivery and breastfeeding experience. In order to ensure homogeneity in the groups, mothers were stratified as mode of delivery (Normal-Cesarean) and breastfeeding experience (Present-Non-existent). After the blocks were formed, the groups included in the study were randomly assigned to the strata with the letters A, B and C using the random numbers table obtained in the computer environment (www.random.org). Which letter would be in which group was determined by lot (A=Odor Stimulation, B=Odor+Taste Stimulation, C=Control Group).
Who Masked: Investigator
Masking Description: According to the a priori power analysis with a pairwise hypothesis, effect size of 0.409, significance level of 0.05 and power of 0.80; it was determined that the inclusion of a total of 72 newborns (Odor Stimulation: 24, Odor+taste stimulation: 24, Control: 24) in the study would provide sufficient sample size.
  Inclusion Criteria; For the mother;
  * Having a term and healthy baby,
  * No communication and language problems,
  * No maternal illness preventing breastfeeding (active chemotherapy, HIV positive, neurological or psychological problems, etc.),
  * Willingness to breastfeed, For the baby;
  * Not having a disease condition that prevents breastfeeding (cleft palate, cleft lip, galactotemia, choanal atresia, etc.),
  * Being at normal birth weight (2500gr-4000gr),
  * Apgar score of 7 and above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Odor stimulation group (Experimental): In the breast milk odor stimulation group, one or two drops of breast milk were placed on a sponge in accordance with the literature. Breast milk was obtained from each infant's own mother by hand expressing. The mothers were asked to express two drops of breast milk from their breasts onto the sponge. The sponge on which the breast milk was dripped was placed as close to the baby's nose as possible without touching the baby's nose. Since breast milk odor stimulation is recommended to be given to the baby for 1 minute in the literature, the baby was allowed to smell the odor of breast milk for 1 minute. The baby was then given to the mother for breastfeeding and breastfeeding was initiated as in routine practice.
  Interventions: Behavioral: Breast Milk Odor Stimulation
- Odor + Taste Stimulation Group (Experimental): In this group in which the breast milk sniffing method was applied; two drops of breast milk were dripped onto a sponge in accordance with the literature and this sponge was placed as close to the nose as possible without touching the nose and the baby was allowed to smell the smell of breast milk for about 1 minute. Then the baby was given to the mother. The mother was asked to express milk manually and to apply/drip approximately 0.2 ml (approximately two drops) of the expressed colostrum starting from the tip of the baby's tongue, along the tongue surface, on both cheeks of the baby, as applied in studies using oral colostrum as a reference. The mother was also asked to express a drop of milk from her breast and manually apply it to the areola. Breastfeeding was then initiated as in routine practice.
  Interventions: Behavioral: Stimulation of Breast Milk Smell and Taste
- Control Group (No Intervention): The control group did not receive any intervention other than the routine initiation of breastfeeding at the clinic. They were provided with breastfeeding education by the lactation counselor.

INTERVENTIONS:
Behavioral: Breast Milk Odor Stimulation — In the breast milk odor stimulation group, one or two drops of breast milk were placed on a sponge in accordance with the literature. Breast milk was obtained from each infant's own mother by hand expressing. The mothers were asked to express two drops of breast milk from their breasts onto the sponge. The sponge on which the breast milk was dripped was placed as close to the baby's nose as possible without touching the baby's nose. Since breast milk odor stimulation is recommended to be given to the baby for 1 minute in the literature, the baby was allowed to smell the odor of breast milk for 1 minute. The baby was then given to the mother for breastfeeding and breastfeeding was initiated as in routine practice.
  Arms: Odor stimulation group
Behavioral: Stimulation of Breast Milk Smell and Taste — In this group in which the breast milk sniffing method was applied; two drops of breast milk were dripped onto a sponge in accordance with the literature and this sponge was placed as close to the nose as possible without touching the nose and the baby was allowed to smell the smell of breast milk for about 1 minute. Then the baby was given to the mother. The mother was asked to express milk manually and to apply/drip approximately 0.2 ml (approximately two drops) of the expressed colostrum starting from the tip of the baby's tongue, along the tongue surface, on both cheeks of the baby, as applied in studies using oral colostrum as a reference. The mother was also asked to express a drop of milk from her breast and manually apply it to the areola. Breastfeeding was then initiated as in routine practice.
  Arms: Odor + Taste Stimulation Group

SUMMARY:
The study aimed to investigate the effects of breast milk sniffing and breast milk tasting and sniffing on sucking success and early feeding cues in term newborns who were started to breastfeed for the first time.

DETAILED DESCRIPTION:
In the literature, there are many studies examining the odor effect or odor and taste effect during gavage feeding of premature and low birth weight infants hospitalized in the Neonatal Intensive Care Unit (NICU). However, no study was found to examine the effect of smell and taste application on breastfeeding success and early feeding cues during initiation of breastfeeding for the first time in healthy term newborns. It is clear that sick newborns need much more support and intervention in the transition to oral feeding. However, the low rates of breastfeeding in our country indicate that the use of effective and facilitating methods to initiate and maintain breastfeeding is also necessary for term and healthy infants. Therefore, this study may guide healthcare professionals on the effectiveness of odor and taste stimulation for early breastfeeding and provide ideas for designing new research and projects.

ELIGIBILITY:
Inclusion Criteria:

* For the mother
* Having a term and healthy baby,
* No communication and language problems,
* No maternal illness preventing breastfeeding (active chemotherapy, HIV positive, neurological or psychological problems, etc.),
* Willingness to breastfeed, For the baby;
* Not having a disease condition that prevents breastfeeding (cleft palate, cleft lip, galactotemia, choanal atresia, etc.),
* Being at normal birth weight (2500gr-4000gr),
* Apgar score of 7 and above.

Exclusion Criteria:

* Under 18 and over 40 years of age,
* Development of postpartum complications (in mother or baby),
* Multiple pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Breastfeeding mothers
Enrollment: 72 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | First measurement-First day of hospitalization
  This form was created by the researchers by utilizing the literature. The descriptive information form consisted of a total of 12 questions inquiring about the mother's descriptive information (maternal age, education level, occupation, place of residence, economic status), obstetric information (mode of delivery, number of deliveries, breastfeeding experience, time of first breastfeeding) and infant information (infant's gender, birth weight, gestational week, Apgar score at 5 min).
Early Feeding Tips Scale | First measurement-first breastfeeding of the first day
  The Turkish validity and reliability study of the scale developed by Thoyre, Ahaker, and Pridham in 2005 was conducted by Girgin et al. in 2021. The early feeding cues scale consists of 19 items and 5 subcategories and is evaluated based on observation. These categories are respiratory regulation, oral-motor function, swallowing coordination, alertness-energy status and physiological stability.The lowest total score is 19 and the highest is 57. A higher score indicates the presence of early feeding cues and a lower score indicates a decrease in early feeding cues.
Breastfeeding Identification and Assessment Scale (LATCH) | First measurement-first breastfeeding of the first day
  It is a measurement tool developed by Jansen and Wallece in 1993, which is similar to the APGAR scoring system in terms of scoring. Turkish validity and reliability studies of the LATCH breastfeeding diagnosis form were conducted by Demirhan in 1997 , Koyun in 2001 , and Yenal and Okumuş in 2003. Each criterion in the scale is given a score between 0 and 2 and the lowest score is 0 and the highest score is 10. An increase in the scores obtained from the scale indicates breastfeeding success.
Early Feeding Tips Scale | Second measurement-Second breastfeeding of the first day
  The Turkish validity and reliability study of the scale developed by Thoyre, Ahaker, and Pridham in 2005 was conducted by Girgin et al. in 2021. The early feeding cues scale consists of 19 items and 5 subcategories and is evaluated based on observation. These categories are respiratory regulation, oral-motor function, swallowing coordination, alertness-energy status and physiological stability.The lowest total score is 19 and the highest is 57. A higher score indicates the presence of early feeding cues and a lower score indicates a decrease in early feeding cues.
Breastfeeding Identification and Assessment Scale (LATCH) | Second measurement-Second breastfeeding of the first day
  It is a measurement tool developed by Jansen and Wallece in 1993, which is similar to the APGAR scoring system in terms of scoring. Turkish validity and reliability studies of the LATCH breastfeeding diagnosis form were conducted by Demirhan in 1997 , Koyun in 2001 , and Yenal and Okumuş in 2003. Each criterion in the scale is given a score between 0 and 2 and the lowest score is 0 and the highest score is 10. An increase in the scores obtained from the scale indicates breastfeeding success.
Early Feeding Tips Scale | Third measurement-Third breastfeeding of the first day
  The Turkish validity and reliability study of the scale developed by Thoyre, Ahaker, and Pridham in 2005 was conducted by Girgin et al. in 2021. The early feeding cues scale consists of 19 items and 5 subcategories and is evaluated based on observation. These categories are respiratory regulation, oral-motor function, swallowing coordination, alertness-energy status and physiological stability.The lowest total score is 19 and the highest is 57. A higher score indicates the presence of early feeding cues and a lower score indicates a decrease in early feeding cues.
Breastfeeding Identification and Assessment Scale (LATCH) | Third measurement-Third breastfeeding of the first day
  It is a measurement tool developed by Jansen and Wallece in 1993, which is similar to the APGAR scoring system in terms of scoring. Turkish validity and reliability studies of the LATCH breastfeeding diagnosis form were conducted by Demirhan in 1997, Koyun in 2001, and Yenal and Okumuş in 2003. Each criterion in the scale is given a score between 0 and 2 and the lowest score is 0 and the highest score is 10. An increase in the scores obtained from the scale indicates breastfeeding success.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Kucukoglu, Study Director — Selcuk University
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published

REFERENCES:
- [Background] Varendi H, Porter RH. Breast odour as the only maternal stimulus elicits crawling towards the odour source. Acta Paediatr. 2001 Apr;90(4):372-5. PMID 11332925
- [Background] Raimbault C, Saliba E, Porter RH. The effect of the odour of mother's milk on breastfeeding behaviour of premature neonates. Acta Paediatr. 2007 Mar;96(3):368-71. doi: 10.1111/j.1651-2227.2007.00114.x. PMID 17407458
- [Background] Yildiz A, Arikan D, Gozum S, Tastekin A, Budancamanak I. The effect of the odor of breast milk on the time needed for transition from gavage to total oral feeding in preterm infants. J Nurs Scholarsh. 2011 Sep;43(3):265-73. doi: 10.1111/j.1547-5069.2011.01410.x. Epub 2011 Jul 25. PMID 21884372
- [Background] Thoyre SM, Shaker CS, Pridham KF. The early feeding skills assessment for preterm infants. Neonatal Netw. 2005 May-Jun;24(3):7-16. doi: 10.1891/0730-0832.24.3.7. PMID 15960007
- [Background] Aykanat Girgin B, Gozen D, Uslubas R, Bilgin L. The Evaluation of Oral Feeding in Preterm Infants: Turkish Validation of the Early Feeding Skills Assessment Tool. Turk Arch Pediatr. 2021 Sep;56(5):440-446. doi: 10.5152/TurkArchPediatr.2021.21008. PMID 35110111
- [Background] Jensen D, Wallace S, Kelsay P. LATCH: a breastfeeding charting system and documentation tool. J Obstet Gynecol Neonatal Nurs. 1994 Jan;23(1):27-32. doi: 10.1111/j.1552-6909.1994.tb01847.x. PMID 8176525